CLINICAL TRIAL: NCT05399836
Title: Subjective Social Status and the Effect of Portion Size Reduction: a 1-day Dietary Behaviour Experimental Study
Brief Title: SSS and the Impact of Portion Size on Daily Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: European Research Council (Other)
Responsible Party: Principal Investigator, Eric Robinson, Principal Investigator (Professor in Psychological Sciences), University of Liverpool
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 803194 SSS PSE
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Diet, Healthy; Eating Behavior; Obesity
Keywords: portion size; socio-economic position; eating behaviour
MeSH Terms: conditions — Feeding Behavior; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Larger portions (Experimental): the main meal component (lunch/dinner) served to participants in the laboratory, reflecting 100% portion. All other foods are identical across conditions (e.g. sides, seconds, dessert, snacks).
  Interventions: Behavioral: Portion size manipulation
- Smaller portions (Experimental): the main meal component (lunch/dinner) served to participants in the laboratory, reflecting 66% portion (i.e. reduced portion size). All other foods are identical across conditions (e.g. sides, seconds, dessert, snacks).
  Interventions: Behavioral: Portion size manipulation

INTERVENTIONS:
Behavioral: Portion size manipulation — The intervention will be administered via changing portion sizes of foods served to participants.

SUMMARY:
Reducing food portion size is a potential strategy to reduce energy intake. However, it remains unclear who is most susceptible to the portion size effect (PSE). There are just two studies which have examined the PSE in the context of socioeconomic position (SEP), with mixed findings. In an online trial the PSE on intended consumption of unhealthy snacks was 18-24% larger for participants of lower SEP compared to participants of higher SEP. However, in a recent laboratory study which examined the PSE on total daily energy intake, participants of lower SEP were no more susceptible to the influence of portion size on eating behaviour than participants of higher SEP. Further research is required to elucidate these divergent findings.

There is also an absence of evidence examining the moderating role of subjective social status (SSS) - an individual's perceived standing in society - on the PSE. Given evidence that the subjective experience of social class may be associated with health outcomes, the present study examines whether reductions to the portion size reduces daily energy intake, and whether and how SSS (higher vs lower) moderates the PSE.

In a crossover experiment, participants will be served all meals in the lab on two separate days, with the portion size of main components at breakfast, lunch and dinner manipulated (i.e. smaller on one day vs larger on the other day). All other foods offered are identical. Food intake from the portion-manipulated breakfast, lunch and dinner, as well as all other meal components (non-portion-manipulated sides, dessert, seconds, snacks, etc.) will be measured, to assess total daily energy intake (kcal).

DETAILED DESCRIPTION:
See Study Protocol attached.

ELIGIBILITY:
Inclusion Criteria:

* Female
* UK (United Kingdom) residents, able to visit laboratory in Liverpool
* Aged 18 or over
* Fluent in English
* willing to consume the test foods
* Self report willingness to eat test foods
* BMI between 18.5 - 32.5kg2

Exclusion Criteria:

* participation in our previous study
* food allergies, intolerances or specific dietary requirements (except vegetarian)
* taking medication which affects appetite
* currently pregnant
* history of eating disorders
* currently on a diet to lose weight

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as female
Enrollment: 47 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Daily energy intake | Time Frame: 24 hours after intervention administered
  Total energy (kcal) consumed from breakfast, lunch, dinner, dessert, snackbox, and any self-reported additional foods.

SECONDARY OUTCOMES:
Energy intake from portion-manipulated foods | Time Frame: 24 hours after intervention administered
  Total energy (kcal) consumed from portion-manipulated foods at breakfast, lunch, and dinner
Energy intake from non portion-manipulated foods | Time Frame: 24 hours after intervention administered
  Total energy (kcal) consumed from other foods (no portion-manipulation) at breakfast, lunch, dinner, snacks, and self-reported foods.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Robinson, PhD, Principal Investigator — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study data (anonymised) will be shared on the Open Science Framework (OSF)
Supporting Information: Study Protocol, SAP
Time Frame: On publication, indefinitely
Access Criteria: Open website
URL: https://osf.io/hx75k/

REFERENCES:
- [Derived] Langfield T, Clarke K, Marty L, Jones A, Robinson E. Socioeconomic position and the influence of food portion size on daily energy intake in adult females: two randomized controlled trials. Int J Behav Nutr Phys Act. 2023 Apr 27;20(1):53. doi: 10.1186/s12966-023-01453-x. PMID 37101143
- Available data/document: Study Protocol — https://osf.io/hx75k/ — Protocol on the Open Science Framework (OSF)
- Available data/document: Statistical Analysis Plan — https://osf.io/hx75k/
- Available data/document: Individual Participant Data Set — https://osf.io/hx75k/ — The study protocol and statistical analysis plan were pre-registered on the OSF prior to starting recruitment. Participant dataset (anonymised) will be made available when results are published.